CLINICAL TRIAL: NCT05277987
Title: A Single Arm, Open Lable and Single Site Early Phase I Clinical Trial to Evaluate the Safety, Cell Kinetics and Initial Efficacy About Anti-claudin18.2 the Specificity of Chimeric Antigen Receptor T Cells in the Advanced Gastric / Esophagogastric Junction Adenocarcinoma and Pancreatic Cancer Subjects
Brief Title: An Evaluation Trial About Anti-claudin18.2 the Specificity of Chimeric Antigen Receptor T Cells in the Advanced Gastric / Esophagogastric Junction Adenocarcinoma and Pancreatic Cancer Subjects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Fifth People's Hospital (Other)
Responsible Party: Principal Investigator, LiuTao, Principal Investigator, Shenzhen Fifth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC-016-GC/PC-101
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: CAR T-Cell Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEC-016 (Experimental): Anti-claudin18.2 the Specificity of Chimeric Antigen Receptor T Cells
  Interventions: Drug: HEC-016(0.5×10^6 CAR-T Cells); Drug: HEC-016(0.5×10^6.5 CAR-T Cells); Drug: HEC-016(0.5×10^7 CAR-T Cells)

INTERVENTIONS:
Drug: HEC-016(0.5×10^6 CAR-T Cells) — The initial dose is set to 0.5 × 10^6 car-t cells / kg, and 3 ~ 6 subjects are expected to be included in the dose group. DLT was observed within 28 days after cell infusion.
Drug: HEC-016(0.5×10^6.5 CAR-T Cells) — The Second dose is set 0.5 × 10^6.5 car-t cells / kg, and 3 ~ 6 subjects are expected to be included in the dose group.
Drug: HEC-016(0.5×10^7 CAR-T Cells) — The Third dose is set 0.5 × 10^7 car-t cells / kg, and 3 ~ 6 subjects are expected to be included in the dose group.

SUMMARY:
An Evaluation Trial About Anti-claudin18.2 the Specificity of Chimeric Antigen Receptor T Cells in the Advanced Gastric / Esophagogastric Junction Adenocarcinoma and Pancreatic Cancer Subjects. To evaluate the tolerability and safety of different doses of HEC-016 CAR-T cell injections in patients with advanced gastric / esophagogastric junction adenocarcinoma and pancreatic cancer, to observe dose limiting toxicity (DLT), to determine the maximum tolerated dose (MTD) and to recommend the regimen for subsequent clinical trials.

DETAILED DESCRIPTION:
Single Site, single arm and open label design are adopted. The dose increment is based on the traditional "3 + 3" method, and the initial dose is set to 0.5 × 10^6 car-t cells / kg, and 3 ~ 6 subjects are expected to be included in each dose group. DLT was observed within 28 days after infusion. One suject of each dose group was enrolled first, and there was no DLT within 14 days before entering the next subject. If the subject had DLT within 14 days, the investigator can evaluate whether the dose group continued to be enrolled and the time interval of the next subject. After completing the safety observation of 3 subjects who meet the DLT evaluation and analysis set in each dose group, they can be increased to the next dose when there is no DLT; If one subject in the first three cases has DLT, another three subjects need to be selected into the dose group (but the researcher can also decide whether to continue to be selected into the dose group according to the actual situation of the subjects). In the process of dose increase, if DLT occurs in ≥ 2 / 3 or ≥ 2 / 6 subjects in a dose group, the dose increase stops.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 70, regardless of gender;
* Subjects with pathologically confirmed advanced gastric / esophagogastric junction adenocarcinoma who failed or did not tolerate at least second-line treatment; Or patients with advanced pancreatic cancer confirmed by pathology, and at least first-line treatment failed or intolerance.
* The immunohistochemical (IHC) staining of tumor tissue samples of the subjects was positive for claudin 18.2 (positive was defined as the positive expression of claudin 18.2 in ≥ 1% of tumor cells detected by IHC in the laboratory; the subjects with adenocarcinoma at the junction of stomach / esophagus and stomach needed HER2 to be negative);
* ECOG score: 0 ~ 2 points
* Expected survival time ≥ 12 weeks;
* According to the solid tumor efficacy evaluation standard (RECIST) v1.1Measurable lesions;
* The functional level of important organs must meet the following requirements (not treated with blood products or hematopoietic growth factors, such as granulocyte colony stimulating factor, erythropoietin, etc. within 2 weeks before screening):

  1. Neutrophil absolute value (ANC) ≥ 1.0 × 10^9/L
  2. Lymphocyte absolute value (ALC) ≥ 0.3 × 10^9/L
  3. Platelet (PLT) ≥ 50 × 10^9/L
  4. Hemoglobin (Hgb) ≥ 70 g / L
  5. International normalized ratio (INR) and activated partial thromboplastin time (APTT) < 1.5 ULN
  6. Serum total bilirubin (TBIL) ≤ 1.5 × ULN (TBIL ≤ 3 for Gilbert syndrome subjects) × ULN）； ALT and AST ≤ 2.5 × ALT and AST ≤ 5, if there is liver metastasis × ULN）
  7. Creatinine clearance calculated according to Cockcroft Gault formula ≥ 50 ml / min
  8. Subjects whose urine routine shows urinary protein ≥ + + should receive 24-hour quantitative detection of urinary protein, and the test result is < 1.0 G
  9. Blood oxygen saturation ≥ 95% in non oxygen absorption state
* Female subjects with fertility: non lactation, blood pregnancy test during screening period must be negative for pregnancy, and they agree to take efficient contraceptive measures during treatment and within 6 months after the last infusion of study treatment; Male subjects who were not sterilized: agreed to take effective contraceptive measures during treatment and within 6 months after the last infusion of study treatment;
* The subjects volunteered to participate in the study and signed a written informed consent by themselves or their guardian.

Exclusion Criteria:

* Previous treatment history in any of the following situations:

  1. Subjects who had received other chemotherapy (except pretreatment chemotherapy and bridging therapy specified in the protocol), small molecule targeted therapy, immunoantitumor therapy (Immune checkpoint inhibitor, etc.), radiotherapy and major surgery within 4 weeks before the first infusion;
  2. Within 4 weeks before the first infusion, received anti-tumor traditional Chinese medicine (with anti-tumor indications approved by nmpa);
  3. Those who receive live vaccine (including attenuated live vaccine) within 4 weeks before the first infusion and / or plan to receive live vaccine after enrollment;
  4. Participated in any intervention clinical trial within 4 weeks before the first infusion (except for the overall survival follow-up subjects participating in a study);
  5. Previously received any cellular immunotherapy (including but not limited to car-t, CIK, NK cell therapy, etc.);
  6. Those who have previously received any targeted therapy for claudin 18.2;
  7. Patients with a history of organ transplantation or allogeneic bone marrow transplantation;
* Not recovered from the adverse reactions of previous anti-tumor treatment (i.e. recovered to ≤ level 1 or baseline level according to CTCAE V5.0);
* Central nervous system metastases currently in need of treatment or uncontrolled central nervous system metastases; Or central nervous system metastasis is confirmed, but it is not stable after anti-tumor treatment for more than 4 weeks (definition of central nervous system metastasis stability: no new neurological defect caused by central nervous system metastasis is found, no new lesions are found in central nervous system imaging examination, and corticosteroid / steroid treatment is not required); Spinal cord compression, cancerous meningitis or leptomeningeal disease;
* In the first 5 years before the first infusion, other malignant tumors except gastric or esophagogastric junction adenocarcinoma or pancreatic cancer were combined. Excluding: tumors with negligible risk of metastasis or death (e.g. expected 5-year OS > 90%) and expected to be curable after treatment (e.g. cervical carcinoma in situ, skin basal cell carcinoma or squamous cell carcinoma, localized prostate cancer treated with radical surgery, breast ductal carcinoma in situ treated with radical surgery), Or any other tumor that has been cured (no evidence of disease recurrence within 5 years);
* Subjects who had thrombosis or embolism events within 12 months before the first infusion, such as cerebrovascular accident (including transient ischemic attack, except lacunar infarction), deep venous thrombosis, pulmonary embolism, etc., or who were receiving thrombolytic or anticoagulant therapy such as warfarin, heparin or other similar drugs
* Massive pleural / ascitic fluid or pericardial effusion with clinical symptoms or requiring symptomatic treatment (puncture or drainage once a month or more frequently);
* The investigator assessed that there is a high risk of unexplained anemia or gastrointestinal bleeding and perforation; Or those who have gastrointestinal bleeding in recent 3 months, including a history of hematemesis, bloody stool or black stool within 3 months; Fecal occult blood (+) and above; Those with occult blood (+) or "positive", "weak positive" or "fecal occult blood transferrin positive" or "fecal occult blood hemoglobin positive" and the primary focus of gastric tumor has not been surgically removed need gastroscopy, and gastrointestinal bleeding may occur according to the judgment of the researcher
* Any past or current active autoimmune disease or history of autoimmune disease, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome (granulomatosis of polyangitis), immune hypophysitis, autoimmune hepatitis, systemic sclerosis (scleroderma, etc.) Hashimoto's thyroiditis (see below for exceptions), autoimmune vasculitis, autoimmune neuropathy (Guillain Barre syndrome), etc. Except for the following cases: type I diabetes, hormone replacement therapy, hypothyroidism (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo without systemic treatment;
* Those who have a history of psychotropic substance abuse and can not quit or have mental disorders;
* Researchers believe that those who have other serious acute or chronic diseases and are not suitable to participate in the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
DLT | Within 28 days after the first infusion
  Dose limiting toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Luohu Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided